CLINICAL TRIAL: NCT07116148
Title: Investigation of a Hybrid Environmental Enrichment-Based Early Intervention Approach for Infants at Risk of Cerebral Palsy
Brief Title: Hybrid Early Intervention for Infants at Risk of Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Izgi Miray Demirbag, Physiotherapist, Medipol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E-10840098-202.3.02-4232
Record Dates: First submitted 2025-07-07; First posted 2025-08-11 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy (CP)
Keywords: Environmental enrichment, early intervention, hybrid model, plasticity, cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The study utilized HEP (Homeostasis Environmental Enrichment Plasticity), an environmental enrichment-based early intervention approach implemented with a hybrid model. The HEP approach is an ecological model that aims to provide multidimensional support to infants at developmental risk during the early developmental period. This approach is based on a holistic synthesis of the biological basis of development and environmental interactions. The intervention is built on a theoretical framework that supports physiological homeostasis, encourages environmental exploration, and activates neuroplasticity. The HEP approach aims to optimize the developmental potential of infants at risk for developmental difficulties through early environmental enrichment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infants at risk of cerebral palsy (Other): The HEP Approach utilizes key principles of enriched environment models and brain plasticity. The therapists and family collaborate during the intervention process to offer permanent, ongoing, personal ized environmental stimulation to promote the child's active exploration and participation. Acrucial component of the HEP Approach is enhancing parenting self-efficacy to create en riched environmental conditions in the home and on an ongoing basis across environments.
  Interventions: Other: The Homeostasis-Enrichment-Plasticity (HEP®) Approach

INTERVENTIONS:
Other: The Homeostasis-Enrichment-Plasticity (HEP®) Approach — The HEPApproach intervention and clinical reasoning process follow a systematic order based on the data-driven decision-making model. There are 11 phases to the HEP Approach process. Phase 1 involves referral to the program. Phase 2 includes a meeting with the family to introduce them to the HEP Approach. Phase 3 is a comprehensive assessment of the child and family systems. Phase 4 is the identification of family and child strengths and challenges based on the assessment. Phase 5 involves formulating hypotheses about how underlying factors or systems impact the child's challenge areas. Phases 6 and 7 include collaborative goal setting and outcome measure identification with the family. Phase 8 is intervention planning. Phase 9 implements the intervention through an individualized process that generally involves four steps that prioritize different areas of need (e.g., self-regulation and homeostasis of the child, adaptation of the physical and social home environment to support succes

SUMMARY:
This study aimed to evaluate the feasibility, safety, and caregiver acceptance of the Homeostasis-Enrichment-Plasticity (HEP®) Approach, a novel early intervention based on the environmental enrichment paradigm, applied as a hybrid model for infants at risk for cerebral palsy (CP). The effects on functional goals, development, and parental well-being will be examined. The intervention consists of weekly one-hour sessions for 12 weeks with 17 infants aged 4-10 months at risk for CP, identified via the Prechtl Assessment or brain imaging. Feasibility and acceptance will be assessed by a 24-item Likert scale. Developmental outcomes will be measured with GAS, Bayley-III, ISFT, and DASS-21.

DETAILED DESCRIPTION:
This study aimed to evaluate the feasibility, safety, caregiver acceptability, and satisfaction levels of the Homeostasis-Enrichment-Plasticity (HEP®) Approach, a novel early intervention model based on the environmental enrichment (EN) paradigm and widely used in the literature, as a hybrid approach for infants at risk for cerebral palsy (CP). Furthermore, the effects of the intervention on the achievement of individualized functional goals, developmental outcomes, and parental well-being will be examined. Unlike previous studies, the HEP intervention in this study will be implemented as a hybrid model, implemented both in the clinic and at home. The intervention will be delivered in one-hour sessions per week for 12 weeks to 17 infants aged 4-10 months corrected age, identified as at risk for CP through either the Prechtl Assessment of General Movements or abnormal brain imaging confirmed by a pediatric neurologist. The feasibility, safety, and caregiver acceptance of the intervention will be assessed using a 24-item Likert-type scale developed by the researcher. Developmental outcomes will be measured by the Goal Attainment Scale (GAS), Bayley Developmental Scales for Infants and Toddlers-III (Bayley-III), Infant Sensory Function Test (ISFT), and Depression Anxiety Stress Scale-21 (DASS-21).

ELIGIBILITY:
Inclusion Criteria:

Infants who meet the following criteria will be included in the study:

* According to the general movement assessment, babies from birth to the 8th week have poor repertoire, synchronized cramps or chaotic movement pattern, and the presence of abnormal fidgeting movements between the 6th and 9th weeks.
* A neurologist has detected the presence of abnormal brain imaging on magnetic resonance imaging or cranial ultrasound,
* Absence of congenital anomalies,
* The family agrees to participate regularly in the study.

Exclusion Criteria:

* Major vision or hearing problems,
* Presence of any genetic syndrome or congenital anomaly,
* Medical conditions that prevent active participation in the study (such as oxygen dependence),
* Participation in other experimental rehabilitation studies

Ages: 4 Months to 10 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility Questionnaire | From July 2025 to November 2025
  A 24-item Likert-type questionnaire was developed by the researcher to evaluate the feasibility, acceptability, satisfaction level, and safety of the intervention. The questionnaire items were grouped under four main categories: feasibility (items 1-7), acceptability (items 8-12), satisfaction (items 13-19), and safety (items 20-24). The five-point Likert-type scale included response options ranging from 1 (Strongly Disagree) to 5 (Strongly Agree).

OTHER OUTCOMES:
Goal Attainment Scaling | From July 2025 to November 2025
  Goal Attainment Scaling (GAS) is one of the most frequently recommended goal-setting methods used in clinical and research settings to measure changes that occur during and after an intervention. Research has shown that GAS is a reliable tool for children with developmental challenges.
  GAS is a scale used to evaluate the extent to which individually set goals-established at the beginning of the intervention-are achieved, providing subjective information related to the infant's specific needs. The scale uses a five-point rating system ranging from -2 to +2 to score goal attainment. A score of 0 represents the expected level of performance; -1 indicates slightly below expectations, and -2 indicates much lower than expected. Similarly, +1 reflects slightly above expectations, and +2 represents much better than expected performance. The scores are converted into standardized scores for analysis, and T-scores are used as outcome measures for the targeted goals.
Bayley Scales of Infant and Toddler Development - Third Edition (Bayley-III) | From July 2025 to November 2025
  The Bayley-III is a widely used tool for assessing the developmental functioning of children between the ages of 1 and 42 months. Its primary purposes are to identify developmental delays, provide professionals with information about a child's strengths and areas in need of support when developing comprehensive intervention plans, and offer a systematic method for monitoring developmental progress.
  The Bayley-III evaluates development across five domains: cognitive, language, motor, social-emotional, and adaptive behavior. The cognitive, language, and motor domains are assessed through direct testing with the child, while the social-emotional and adaptive behavior domains are evaluated through questionnaires completed by the caregiver.
Test of Sensory Functions in Infants | From July 2025 to November 2025
  The test consists of five subdomains: response to deep pressure touch, adaptive motor functions, visual-tactile integration, oculo-motor control, and response to vestibular stimulation. It includes a total of 24 items.
  In the response to deep pressure touch subdomain, the infant's reactions to tactile stimuli applied to the arms, hands, abdomen, soles of the feet, mouth, and shoulders are assessed. Responses are scored as 0 (aversive), 1 (mildly defensive), or 2 (integrated).
  The adaptive motor response subdomain evaluates the infant's motor planning ability and the skill to explore various objects with the hands. Scores range from 0 (no response), 1 (disorganized), 2 (partial), to 3 (organized).
  In the visual-tactile integration subdomain, the infant's responses to objects placed on or touching the body are assessed. Scoring is as follows: 0 (hyperresponsive), 1 (hyporesponsive), 2 (normal).
  The oculo-motor control subdomain examines visual tracking and lateralization of the eyes
Depression Anxiety Stress Scales-21 (DASS-21) | From July 2025 to November 2025
  The DASS-21 is a validated and reliable tool for screening depressive and anxiety disorders, and it effectively assesses the severity of three psychological states through 21 items. The scale consists of three subscales: depression (7 items), anxiety (7 items), and stress (7 items). Each item is rated on a 4-point Likert scale ranging from 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time). Lower scores on the subscales indicate better psychological well-being.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Sense On, Ltd., Istanbul, Beykoz
  - Sense On, Istanbul, Beykoz